CLINICAL TRIAL: NCT01467830
Title: Open Inguinal Hernia Repair With Mesh,the Use of Absorbable Versus Non Absorbable Fixation Sutures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: absorbable suturesCTIL
Record Dates: First submitted 2011-10-30; First posted 2011-11-09 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2011-12

CONDITIONS: Inguinal Hernia
Keywords: absorbable sutures efficacy; reducing Adverse effect to be caused from surgery; Inguinal Hernia repair with mesh
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- absorbable sutures (Experimental): patients attributed to that arm, undergoing surgery of Open Inguinal Hernia Repair With Mesh Fixation using absorbable sutures.
  Interventions: Procedure: Open Inguinal Hernia Repair With Mesh,the Use of Absorbable Versus Non Absorbable Fixation Sutures
- non absorbable sutures (Other): patients attributed to that arm, undergoing surgery of Open Inguinal Hernia Repair With Mesh Fixation using non absorbable sutures,this is the method being considered the standard of care thus far.
  Interventions: Procedure: Open Inguinal Hernia Repair With Mesh,the Use of Absorbable Versus Non Absorbable Fixation Sutures

INTERVENTIONS:
Procedure: Open Inguinal Hernia Repair With Mesh,the Use of Absorbable Versus Non Absorbable Fixation Sutures — use of absorbable sutures to fixate mesh inguinal hernia repair.

SUMMARY:
The purpose of this study is to determine the efficacy of mesh fixation using absorbable versus non-absorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing initial unilateral Open Inguinal Hernia Repair surgery.

Exclusion Criteria:

* patients having repeated Inguinal Hernia or bilateral Hernia
* patients undergoing laparoscopic surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Impact of absorbable sutures in inguinal hernia repair on hernia recurrence and post operative outcome | two years
  Absorbable sutures efficacy will be assessed according to:severity of post surgical pain(using NRS-Numerical Rating Scale measure),hernia recurrence (assessed by physical examination during the follow-up period) and other post surgical complications such as nerve entrapment,hematoma and stich granuloma

CONTACTS AND LOCATIONS:
Overall Officials: Adel Abu_salih, M.D, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel